CLINICAL TRIAL: NCT04099225
Title: Multiple Breath Washout (MBW) Using Sulfur Hexafluoride Reference Values and Influence of Anthropometric Parameters
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Dr. Frederik Trinkmann, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: MBW-normal values
Record Dates: First submitted 2019-09-18; First posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Healthy Subjects; Smokers; Non-smokers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Multiple breath washout (MBW) testing — Lung clearance index (LCI), acinar (Sacin) and conductive (Scond) ventilation heterogeneity were derived from triplicate SF6-MBW measurements. Global ventilation heterogeneity was calculated for the 2.5% (LCI2.5) and 5% (LCI5) stopping points.

SUMMARY:
Multiple breath washout (MBW) using Sulphur hexafluoride (SF6) has the potential to reveal ventilation heterogeneity in obstructive lung disease which is frequent in patients with small airway disease. However, it is missed by commonly used tests with reference data being scarce and mostly restricted to younger collectives. We aimed to evaluate the influence of anthropometric parameters on SF6-MBW reference values in pulmonary healthy adults.

ELIGIBILITY:
Inclusion Criteria:

non-smoker

* no history of pulmonary disease
* absence of dyspnoea, cough, thoracic pain
* no self-reported smoking history
* normal lung function testing

  * normal shape of flow-volume curve
  * normal shape of flow-pressure curve
  * FEV1/FVC >70% (forced expiratory volume in 1 second / forced vital capacity)
  * TLC > 80% of predicted (total lung capacity)
  * TLCO/VA > 80% of predicted (transfer factor corrected for ventilated alveolar volume)
  * R5 < 150% of predicted (resistance at 5Hz, impulse oscillometry)

smoker

- as above, but with self-reported smoking history >10 pack years

Exclusion Criteria:

* unwilling or unable to give informed consent
* history of any respiratory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers including never, active and former smokers
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Lung clearance index (LCI) derived from multiple breath washout testing (MBW) | 30 minutes
  global ventilation heterogeneity

SECONDARY OUTCOMES:
Acinar phase-III-slope (Sacin) derived from multiple breath washout testing (MBW) | 30 minutes
  local ventilation heterogeneity
Conductive phase-III-slope (Scond) derived from multiple breath washout testing (MBW) | 30 minutes
  local ventilation heterogeneity

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Trinkmann, MD, Principal Investigator — University Medical Center Mannheim

IPD SHARING:
Plan to Share IPD: No
Sharing of individual participant data is prohibited by data protection regulations. Summarized data including the models will be made available thru an online repository (GitHub).

REFERENCES:
- [Derived] Trinkmann F, Maros M, Roth K, Hermanns A, Schafer J, Gawlitza J, Saur J, Akin I, Borggrefe M, Herth FJF, Ganslandt T. Multiple breath washout (MBW) testing using sulfur hexafluoride: reference values and influence of anthropometric parameters. Thorax. 2021 Apr;76(4):380-386. doi: 10.1136/thoraxjnl-2020-214717. Epub 2021 Feb 16. PMID 33593931